CLINICAL TRIAL: NCT07128823
Title: Combined Effects of Accelerated Skill Acquisition Programme With Segmental Vibration on Extensor Muscles for Upper Limb Function in Subacute Stroke.
Brief Title: Effects of Accelerated Skill Acquisition Programme With Segmental Vibration on Upper Limb in Stroke.
Acronym: ASAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0259 Mubeen Arshad
Record Dates: First submitted 2025-04-07; First posted 2025-08-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Subacute Stroke
Keywords: Task orientated training; Segmental vibration; Extensor muscles; Accelerated Skill Acquisition Programme

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): (High-frequency segmental vibration and ASAP with with Routine Physical Therapy)
  Interventions: Other: Group A (High-frequency segmental vibration and ASAP with Routine Physical Therapy)
- Group B (Experimental): Accelerated skill acquisition programme with Routine Physical Therapy
  Interventions: Other: Group B (Accelerated Skill Acquisition Programme with Routine Physical Therapy)

INTERVENTIONS:
Other: Group A (High-frequency segmental vibration and ASAP with Routine Physical Therapy) — A Segmental vibration device was used to provide vibratory stimulation with a frequency of 100 Hz and an amplitude of 1.0 mm. This stimulation was used because vibratory stimulation with a high frequency (80-120 Hz) and low amplitude can elicit strong activity in Ia afferents from the muscle spindles. 100 Hz frequency vibration was applied perpendicularly along the muscle fibers of the forearm extensor muscle (extensor carpi ulnaris (ECU), extensor carpi radialis (ECR), triceps).
  The Accelerated Skill Acquisition Programme (ASAP), a structured, taskoriented motor training program for the upper extremities, is a best-practice synthesis implementing neuroscientific evidence regarding motor training approaches and schedules. The Accelerated Skill Acquisition Program (ASAP) for subacute stroke patients focuses on integrating motor training with motivational enhancement and impairment mitigation.
  Arms: Group A
Other: Group B (Accelerated Skill Acquisition Programme with Routine Physical Therapy) — Exercises within the ASAP typically include:
  Task-Specific Training: Patients engage in activities that mimic daily tasks, such as reaching, grasping, and manipulating objects, to improve their functional abilities Repetitive Practice: Patients perform repetitive movements to strengthen neural pathways and improve motor skills. This can involve tasks like buttoning a shirt, picking up small objects, or pouring water Bilateral Arm Training: This approach involves using both arms simultaneously to perform coordinated tasks, enhancing bimanual skills and improving upper extremity functions Motivational Strategies: The program incorporates motivational techniques to enhance patient engagement and adherence to the exercises, ensuring sustained practice and better outcomes.
  Arms: Group B

SUMMARY:
Stroke is a major health burden and the leading cause of serious long-term disability around the world. One of the most cumbersome deficits after a unilateral stroke is impairment in the contralateral upper limb. Segmental vibration is an intervention that incorporates sensory stimulation to improve motor cortical excitability. This study aims to investigate the influence of a 15-minute SMV application along with accelerated skill acquisition programme (ASAP) on spasticity, motor function, manual dexterity, and somatosensory function of the Upper Limb in Subacute stroke.

This study will be a randomized clinical trial conducted in the physiotherapy department of DHQ Hospital Gujranwala, Gondal Hospital, and Dayan Physiotherapy and Rehabilitation over 10 months. Using the Online Randomizer tool, 60 stroke patients will be recruited through a non-probability convenience sampling technique and randomly divided into two equal groups, Group A and Group B. Group A will receive ASAP with high-frequency segmental vibration(100Hz) on the extensor muscles while Group B, will receive accelerated skill acquisition programme (ASAP) with only. The Assessment tools are the Fugl-Meyer Assessment Scale (for upper limb function), Wolf Motor Functional Test(for motor function), Modified Ashworth Scale(for spasticity), Maximal Hand Grip Strength(for manual dexterity), Nottingham Sensory Assessment(for somatosensory function). Outcome measures will be assessed at baseline,4th week,8th week, and 12th week. Follow-up will be performed in the 16th week. Data analysis will be done by SPSS version 28.0. Two-way Mixed ANOVA, repeated measure ANOVA, and one-way ANOVA will be used in case of normal distribution of data. The Friedman, Kruskal Wallis, and Wilcoxon sign rank tests will be used for non-normal data.

DETAILED DESCRIPTION:
A stroke is a clinically defined syndrome of rapidly developing symptoms or signs of focal loss of cerebral function with no apparent cause other than that of vascular origin. Still, the loss of function can at times be global (applied to patients in a deep coma and those with subarachnoid hemorrhage. Stroke affects approximately 80.1 million people worldwide and causes 5.5 million deaths annually. The risk of stroke is highest between the ages of 55 and 65. Impaired functional movement in a paretic hand is a common post-stroke challenge. Upper extremity hemiparesis is one of the most common symptoms after stroke. Approximately 55%-75% of stroke survivors suffer from upper extremity moto dysfunction, 40% experience moderate to severe problems in the upper extremity. Which can have a considerable impact on activities of daily living and ultimately lead to a significant reduction in quality of life. The segmental vibrator with (ASAP) Task-Oriented training may have the potential to offer targeted, precise, and adaptable interventions, possibly optimizing the rehabilitation process by reinforcing the neural pathways associated with specific movements, promoting better improvement of motor tasks, their efficacy will aid in providing the rehabilitation strategies that may optimize the upper limb function in sub-acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke between 3 months and 6 months post-stroke.
* Fugl-Meyer assessment upper extremity (FMA-UE) motor scores between 19 and 58.
* Participants be able to follow the researcher's instructions and study procedures.
* Spasticity of spastic agonist muscles ranging from 0-2 on the modified Ashworth scale
* Montreal Cognitive Assessment (MoCA) score of 24 or higher, indicating sufficient cognitive function to participate in stroke rehabilitation.

Exclusion Criteria:

Patients with acute or chronic neurologic or orthopedic impairments and those who experienced discomfort or had undergone surgery in the upper limbs within 6 months before the study onset. (30)

* Pain (FMA-UE pain score of 1 for at least 2 joints) in the affected UE.(32)
* All types of aphasia.(38)
* Visual problems that could not be corrected.(39)
* Individuals with unstable medical conditions that could interfere with rehabilitation progress or pose risks during therapy sessions are typically excluded(40)
* Patients with uncontrolled psychiatric disorders that could compromise their ability to participate in or benefit from rehabilitation are typically excluded(41)
* Metal implants e. g cardiac pacemaker

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Assessment at baseline, after 4th,8th,12th and 16th weeks
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess the functioning, balance, sensation, and joint functioning in patients with stroke hemiplegia (0-126 points). Higher scores indicate better motor recovery, with subscores for specific domains like upper extremity (0-66).

SECONDARY OUTCOMES:
Wolf Motor Functional Test (WMFT) | Assessment at baseline, after 4th,8th,12th and 16th week
  The Wolf Motor Functional Test (WMFT) measures upper extremity (UE) motor abilities by scoring 15 tasks on performance time and functional ability, with scores ranging from 0 (unable) to 5 (normal). Lower times and higher functional scores indicate better motor recovery.
Modified Ashworth scale (MAS) | Assessment at baseline, after 4th ,8th ,12th and at 16th week.
  The Modified Ashworth Scale (MAS) measures spasticity in stroke patients by assessing muscle resistance to passive movement, scored from 0 to 4. A score of 0 indicates no increase in muscle tone, while 4 denotes a rigid limb. It is widely used in stroke rehabilitation to evaluate spasticity in upper or lower limbs. Higher scores correlate with greater spasticity.
Maximal Hand Grip Strength (MHGS) | Assessment at baseline, after 4th ,8th ,12th and at 16th week.
  Maximal Hand Grip Strength (MHGS) is a key measure of upper limb function in stroke patients, typically assessed using a dynamometer. In subacute stroke, MHGS scores reflect muscle weakness, with values often ranging from 0-30 kg (compared to 40-50 kg in healthy adults), depending on severity. Lower scores indicate greater impairment, correlating with reduced functional ability in tasks like grasping.
Nottingham Sensory Assessment (NSA) | Assessment at baseline, after 4th,8th,12th and 16th week.
  The Nottingham Sensory Assessment (NSA) is a standardized tool to evaluate sensory impairments in stroke patients, focusing on tactile sensation, proprioception, and stereognosis in the upper and lower limbs. It includes 20 items scored on a 3-point scale (0 = absent, 1 = impaired, 2 = normal), with separate testing for affected and unaffected sides. it takes about 15-20 minutes and is reliable for detecting sensory deficits post-stroke.

OTHER OUTCOMES:
MoCA (Montreal Cognitive Assessment) | Assessment at baseline.
  The Montreal Cognitive Assessment (MoCA) is a one-page, 30-point cognitive screening measurement scale that takes about 10 minutes to administer. There are 12 subtasks in the MoCA test that include memory, visuospatial orientation, executive functioning, phonemic fluency, and two-item abstract thinking task, attention, concentration, and working memory, language, orientation to time and place. A score of 26 is a cutoff score to differentiate between normal and abnormal. The reliability of the MoCA-S was 0.89 and the intraclass correlation coefficient was 0.955.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital Gujranwala, Gondal Hospital, and Dayan Physiotherapy and Rehabilitation, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adhikari SP , Gautam M . The Effectiveness of Accelerated Skill Acquisition Program for Upper Extremity Motor Training in Bilateral Stroke. Kathmandu Univ Med J (KUMJ). 2019 Oct.-Dec.;17(68):341-343. PMID 33311046
- [Background] Thant AA, Wanpen S, Nualnetr N, Puntumetakul R, Chatchawan U, Hla KM, Khin MT. Effects of task-oriented training on upper extremity functional performance in patients with sub-acute stroke: a randomized controlled trial. J Phys Ther Sci. 2019 Jan;31(1):82-87. doi: 10.1589/jpts.31.82. Epub 2019 Jan 29. PMID 30774211
- [Background] Moon JH, Cho HY, Hahm SC. Influence of Electrotherapy with Task-Oriented Training on Spasticity, Hand Function, Upper Limb Function, and Activities of Daily Living in Patients with Subacute Stroke: A Double-Blinded, Randomized, Controlled Trial. Healthcare (Basel). 2021 Aug 3;9(8):987. doi: 10.3390/healthcare9080987. PMID 34442124
- [Background] Kimura N, Sato M, Kobayashi Y, Naito E. Augmented activity of the forearm extensor muscles induced by vibratory stimulation of the palm of the hand in individuals with subacute post-stroke hemiplegia. Brain Inj. 2022 May 12;36(6):782-791. doi: 10.1080/02699052.2022.2048694. Epub 2022 Apr 17. PMID 35430945
- [Background] Choi W. The Effect of Task-Oriented Training on Upper-Limb Function, Visual Perception, and Activities of Daily Living in Acute Stroke Patients: A Pilot Study. Int J Environ Res Public Health. 2022 Mar 8;19(6):3186. doi: 10.3390/ijerph19063186. PMID 35328874
- [Background] Abit Kocaman A, Onal B, Sertel M, Karaca G. The effect of local vibration applied to the forearm extensor muscles on hand function and muscle activation in stroke patients: a randomized controlled study. Acta Neurol Belg. 2023 Oct;123(5):1957-1964. doi: 10.1007/s13760-023-02335-6. Epub 2023 Jul 23. PMID 37481756
- [Background] Tavernese E, Paoloni M, Mangone M, Mandic V, Sale P, Franceschini M, Santilli V. Segmental muscle vibration improves reaching movement in patients with chronic stroke. A randomized controlled trial. NeuroRehabilitation. 2013;32(3):591-9. doi: 10.3233/NRE-130881. PMID 23648613
- [Background] Annino G, Alashram AR, Alghwiri AA, Romagnoli C, Messina G, Tancredi V, Padua E, Mercuri NB. Effect of segmental muscle vibration on upper extremity functional ability poststroke: A randomized controlled trial. Medicine (Baltimore). 2019 Feb;98(7):e14444. doi: 10.1097/MD.0000000000014444. PMID 30762754
- [Background] Arya KN, Verma R, Garg RK, Sharma VP, Agarwal M, Aggarwal GG. Meaningful task-specific training (MTST) for stroke rehabilitation: a randomized controlled trial. Top Stroke Rehabil. 2012 May-Jun;19(3):193-211. doi: 10.1310/tsr1903-193. PMID 22668675
- [Background] Caliandro P, Celletti C, Padua L, Minciotti I, Russo G, Granata G, La Torre G, Granieri E, Camerota F. Focal muscle vibration in the treatment of upper limb spasticity: a pilot randomized controlled trial in patients with chronic stroke. Arch Phys Med Rehabil. 2012 Sep;93(9):1656-61. doi: 10.1016/j.apmr.2012.04.002. Epub 2012 Apr 13. PMID 22507444
- [Background] Noma T, Matsumoto S, Shimodozono M, Etoh S, Kawahira K. Anti-spastic effects of the direct application of vibratory stimuli to the spastic muscles of hemiplegic limbs in post-stroke patients: a proof-of-principle study. J Rehabil Med. 2012 Apr;44(4):325-30. doi: 10.2340/16501977-0946. PMID 22402727
- [Background] Anwer S, Waris A, Gilani SO, Iqbal J, Shaikh N, Pujari AN, Niazi IK. Rehabilitation of Upper Limb Motor Impairment in Stroke: A Narrative Review on the Prevalence, Risk Factors, and Economic Statistics of Stroke and State of the Art Therapies. Healthcare (Basel). 2022 Jan 19;10(2):190. doi: 10.3390/healthcare10020190. PMID 35206805
- [Background] GBD 2016 Stroke Collaborators. Global, regional, and national burden of stroke, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):439-458. doi: 10.1016/S1474-4422(19)30034-1. Epub 2019 Mar 11. PMID 30871944